CLINICAL TRIAL: NCT02602106
Title: Effects of Regular Aquatic Activities on Pregnancy Outcomes
Brief Title: Regular Aquatic Activities and Pregnancy Outcomes
Acronym: aquapreg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Ruben Barakat Carballo, PhD in Physical Exercise and Sports Sciences, Universidad Politecnica de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UFLO_UPM_12
Record Dates: First submitted 2015-10-30; First posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Weight Gain
Keywords: Aquatic activities; Aerobic exercise; Resistance exercise; Pregnancy; Maternal weight gain; birthweight
MeSH Terms: conditions — Weight Gain; Gestational Weight Gain; Birth Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): The aquatic exercise program included a total of three 50-55 minutes session per week. Pregnant women started at 9 weeks and finished at 38-39 weeks.
  Each session included 10 minutes of warm up and 10 minutes of cool down including an specific pelvic floor muscle training. The core section of the session included aerobic and strength moderate exercise in water during 25 to 30 minutes
  Interventions: Behavioral: Aquatic activities intervention
- Control group (No Intervention): Sedentary healthy pregnant women

INTERVENTIONS:
Behavioral: Aquatic activities intervention — Women were suggested to exercise regularly through aquatic activities. A professional in physical exercise and sports designed and conducted the aquatic exercise program.
  Arms: Intervention group

SUMMARY:
Aquatic activities is one of the most attractive physical exercise during pregnancy, especially during the third trimester.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effect of moderate regular aquatic exercise during pregnancy on maternal and fetus outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women without any medical or obstetric complication to practice moderate exercise
* Being able to communicate in Spanish

Exclusion Criteria:

* Being interesting in the study after 16 weeks of gestation
* Having obstetric contraindications
* Not attended regular to the exercise program

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Maternal gestational weight gain | 40-42 weeks
  Maternal weight gain was collected at the end of pregnancy as well as before getting pregnant (pre-gestational weight gain)
Birthweight | 37-42 weeks
  Birth weight was collected at delivery

SECONDARY OUTCOMES:
Number of participants with adverse pregnancy outcomes as assessed by medical records | 37-42 weeks
  Other health baby outcomes at delivery
Gestational age | 37-42 weeks
  Gestational age of pregnancy
Maternal blood pressure and gestational diabetes as assessed by medical records | 9 to 42 weeks
  Blood pressure, gestational diabetes...

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Barakat Carballo, PhD, Principal Investigator — Technical University of Madrid
Locations (1):
- Thecnical University of Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Bacchi M, Mottola MF, Perales M, Refoyo I, Barakat R. Aquatic Activities During Pregnancy Prevent Excessive Maternal Weight Gain and Preserve Birth Weight: A Randomized Clinical Trial. Am J Health Promot. 2018 Mar;32(3):729-735. doi: 10.1177/0890117117697520. Epub 2017 Mar 9. PMID 28279085